CLINICAL TRIAL: NCT03381469
Title: Association Between Periodontitis and Adverse Pregnancy Outcomes in Metabolic Syndrome Patients- Interventional Study
Brief Title: Periodontitis and Adverse Pregnancy Outcomes in Metabolic Syndrome Patients- Interventional Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riyadh Colleges of Dentistry and Pharmacy (Other)
Responsible Party: Principal Investigator, Dr. Ghousia Sayeed, Assistant Professor, Riyadh Colleges of Dentistry and Pharmacy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MetS in Pregnancy
Record Dates: First submitted 2017-12-11; First posted 2017-12-22 (Actual); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Low Birth Weight Baby; Metabolic Syndrome; Pregnancy Complications; Adverse Pregnancy Outcomes; Periodontitis; Premature Birth
MeSH Terms: conditions — Metabolic Syndrome; Pregnancy Complications; Periodontitis; Premature Birth

STUDY DESIGN:
Intervention Model Description: Three groups of patients will be examined parallel to each other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Periodontitis patients undergoing NSPT (Experimental): Case group participants will receive comprehensive periodontal treatment also known as non-surgical periodontal therapy (NSPT) that will be completed by the end of week 20-21 of gestation.
  Interventions: Procedure: Comprehensive periodontal treatment
- Periodontitis Patients undergoing supragingival scaling (Active Comparator): The control group participants with periodontitis will receive oral hygiene instruction and single visit supragingival scaling of all teeth at their baseline visit.
  Interventions: Procedure: single visit supragingival scaling
- Without Periodontitis undergoing supragingival scaling (Active Comparator): Placebo group participants without periodontitis will receive oral hygiene instruction and single visit supragingival scaling of all teeth at their baseline visit.
  Interventions: Procedure: single visit supragingival scaling

INTERVENTIONS:
Procedure: Comprehensive periodontal treatment — The Case group participants will receive non-surgical periodontal therapy that will be completed by the end of week 20-21 of gestation. This will consist of oral hygiene instruction with comprehensive periodontal treatment which will include excavation and sealing of cavities, removal of overhanging restorations, extraction of hopeless teeth followed by supragingival and subgingival scaling and root planing (SRP) of sites with PDs > 4 mm and polishing of all the teeth. Participants will be offered treatment under local anesthetic when necessary. No limits will be imposed on the number of dental visits needed to accomplish periodontal therapy.
  Other Names: Non Surgical Periodontal Therapy (NSPT)
  Arms: Periodontitis patients undergoing NSPT
Procedure: single visit supragingival scaling — The control and Placebo group participants will receive oral hygiene instruction and supragingival cleaning of all teeth at their baseline visit.
  Arms: Periodontitis Patients undergoing supragingival scaling; Without Periodontitis undergoing supragingival scaling

SUMMARY:
Aim The Aim of the current study is to establish the association between periodontitis and adverse pregnancy outcomes in metabolic syndrome (Mets) patients and to evaluate the effect of intervention.

Objectives

1. To evaluate the changes in periodontal status of pregnant women with metabolic syndrome after non surgical periodontal therapy (NSPT)
2. To evaluate the inflammatory marker levels in serum of pregnant women with metabolic syndrome after non surgical periodontal therapy
3. To evaluate the effect of NSPT on adverse pregnancy outcomes of women with metabolic syndrome

DETAILED DESCRIPTION:
Research Design/Methodology Ethics approval will be obtained from Institution Review Board of Riyadh Colleges of Dentistry and Pharmacy.

Sample size calculation (Green, 1991) By considering the Green's formula as below; Medium effect size (R2=0.07) variance in dependent variable accounted for by the independent variable. Beta weights of (ß=0.20). N≥104+k (Number of independent variable) .Hence total sample size required by considering 8 independent variables will be N=104+8=112. Expecting a patient drop out rate of 30%, the sample size is being increased to 50 patients per group. Approximately 150 patients will be recruited from maternity hospitals of Riyadh City.

Written informed consent will be obtained from patients after explaining the details of the study. Patients will be evaluated using a detailed questionnaire. Demographic characteristics such as age, diet, medical history etc will be recorded. All participants will be interviewed by principal investigator at each visit to capture oral hygiene knowledge and behaviors and exposure to risk factors for adverse pregnancy outcomes. Reviews of medical records will be conducted by principal investigator to record pregnancy history, document the course of the current pregnancy, and record any adverse events. All patients will be advised to report immediately to our dental clinic in case they have any dental related issues during the study period.

Examination Procedure All dental examinations will be performed by principal investigator. Clinical oral examinations will record number of teeth, the number of filled and carious teeth.

Outcome Measures: Periodontal parameters: Gingival Index, Plaque Index, Bleeding on probing, Probing depth (PD), Clinical attachment loss (CAL)

A complete periodontal examination will be conducted with the following assessments:

Bleeding on probing, Probing depth and clinical attachment level will be evaluated at six sites per tooth, whereas plaque index and gingival index will be evaluated at four sites per tooth.

Gingival index (GI). All teeth except third molars will be evaluated for gingival inﬂammation using a modiﬁcation of the Loe and Silness , 1963 GI. The GI uses the following scores: 0 = normal gingiva; 1 = mild inﬂammation; 2 = moderate inﬂammation; and 3 = severe inﬂammation.

Plaque index (PI). Prebrushing plaque scores for the buccal surface of each tooth will be assigned using a zero to three scale (Silness and Loe, 1964 ) PI, with ''0''indicating an absence of plaque on the clinical crown and a ''3'' indicating the presence of soft deposits covering more than two-thirds of the crown.

Bleeding on probing (BOP). BOP will be assessed during and recorded after probing measures will be taken for each quadrant. The scoring will be as follows:

0 = absence of bleeding; 1 = bleeding present.

Probing depth. and gingival recession .A manual periodontal probe University of North Carolina -15 probe (UNC-15) , Hu-Friedy, Chicago, Illinois ,will be used to record on all teeth present in the mouth.

Probing depth will be calculated from gingival margin to base of pocket. CAL will be calculated using the clinically detectable cemento-enamel junction (CEJ) as reference and it will be measured from CEJ to base of pocket.

Case definition of Periodontitis outlined by Page & Eke (2007) will be used. The case deﬁnition for severe periodontitis requires two or more interproximal sites with CAL > 6 mm, not on the same tooth, and one or more interproximal sites with PD >5 mm. Moderate periodontitis is deﬁned as two or more interproximal sites with CAL >4 mm, not on the same tooth, or two or more interproximal sites with PD >5 mm, not on the same tooth.

Adult Treatment Panel (ATP) III criteria for Mets will be met if an individual has three or more of the following components (Dos Prazeres Tavares et al, 2016):

Abdominal obesity: waist circumference >88 cm (35 inches) in women; Pregestation Body mass index (BMI) > 30kg/m2 High fasting glucose (FPG): serum glucose level > 110 mg/dl (6.1 mmol/l) or on treatment for diabetes; High blood pressure (BP): systolic BP >130 mm Hg and/or diastolic BP >85 mm Hg or on treatment for hypertension (HTN) Hypertriglyceridemia: serum triglyceride level >150 mg/dl (1.69 mmol/l); and Low high-density lipoprotein (HDL) cholesterol: Serum HDL cholesterol <50 mg/dl (1.29 mmol/l) in women.

Clinical data and samples of blood will be collected at three intervals

* At baseline (before 20 weeks gestation)
* 8 weeks after completion of periodontal therapy
* Within 1-2 days of delivery

Serum bio markers: Interleukin-6(IL-6), Prostaglandin-E2 (PG-E2)

Pregnancy Outcomes: Preterm birth < 37 weeks, Low birth weight < 2500 gms, Preterm low birth weight.

The patients and technicians who will perform the lab analyses will be blinded to group assignment.

Study Design It is a randomized clinical trial. Group 1- Case- Periodontitis patients undergoing Comprehensive periodontal treatment Group 2- Control- Periodontitis Patients undergoing single visit supragingival scaling Group 3- Placebo- Patients without Periodontitis undergoing single visit supragingival scaling After the collection of clinical data, the participants will be randomly allocated to either groups of the study using sealed opaque envelopes labeled with a study number and containing the group allocation. Allocations will be computer generated by a third person who will not otherwise be involved in the study. The Case group participants will receive non-surgical periodontal therapy that will be completed by the end of week 20-21 of gestation. This will consist of oral hygiene instruction with comprehensive periodontal treatment which will include excavation and sealing of cavities, removal of overhanging restorations, extraction of hopeless teeth followed by supragingival and subgingival scaling and root planing (SRP) of sites with PDs > 4 mm and polishing of all the teeth. Participants will be offered treatment under local anesthetic when necessary. No limits will be imposed on the number of dental visits needed to accomplish periodontal therapy.

The control and Placebo group participants will receive oral hygiene instruction and supragingival cleaning of all teeth at their baseline visit. Clinical periodontal related data will be collected at a subsequent review appointment 8 weeks after treatment for all groups.

All control participants will be offered the opportunity to attend for comprehensive periodontal therapy postpartum.

Blood samples will be collected after 10 hours of over night fasting. Serum triglyceride, Serum HDL cholesterol and serum glucose will be quantified using standard laboratory procedures in same medical laboratory for all samples collected.

A 5-ml sample of peripheral venous blood will be collected by vein puncture. The blood samples will be centrifuged at 3000 g for 5 min and the serum will be separated. The serum samples will be frozen in plastic vials at -20º Centigrade until further analyzing. Commercially available ELISA assays will be used to measure concentrations of IL-6, and PGE2 in blood samples, according to the manufacturer's recommendations.

Data analysis will be done using Statistical Package for the Social Sciences (SPSS) software. Mean and standard deviation for all clinical parameters. Diﬀerences between groups will be assessed using independent t-tests. Sample distribution according to demographic, socio-economic and behavioral data will be assessed using chi-square and Fisher_s exact tests. Between-group differences on the distribution of obstetric data will be assessed using Fisher_s exact test, and diﬀerences in adverse pregnancy outcomes will be compared using the independent t-test. Serum bio markers will be presented as median and 25% and 75% percentiles. Diﬀerences between groups will be assessed using the Mann- Whitney U-test, and diﬀerences among experimental periods will be assessed using the Wilcoxon signed-rank test. The Holm-Bonferroni method will be used to adjust for multiple comparisons. Statistical signiﬁcance will be set at 5%

ELIGIBILITY:
Inclusion criteria:

* Patients with Mets
* Primi gravida
* Singleton pregnancy < 20 weeks gestation
* 18-34 years of age
* More than 20 teeth in the mouth

Exclusion criteria:

* Previous history of abortion
* Assisted reproduction procedures like fertility medication or in vitro fertilization
* Positive history of HIV
* Positive history of genitourinary infections in previous 6 months
* Any medical contraindication to periodontal probing
* Undergone periodontal treatment or using chlorhexidine or other mouth rinses in the previous 6 months
* Rampant decay
* Taken systemic antibiotic or anti-inﬂammatory drugs in the last 6 months before the start of the study, or reported use of phenytoin, cyclosporine, calcium antagonists and/or hormone replacement therapy
* Alcoholics
* Smokers and ex-smokers
* History of kidney, liver or lung disease
* History of any other chronic or acute infections during the previous 6 months as assessed on clinical examination or routine lab testing

Ages: 18 Years to 34 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female only
Enrollment: 150 (Estimated)
Dates: Start 2018-02-10 (Actual); Primary Completion 2018-08-01 (Estimated); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
Periodontal parameters- Change in Gingival Index | • At baseline (before 20 weeks gestation) • 8 weeks after completion of periodontal therapy • Within 1-2 days of delivery
  Gingival index (GI). All teeth except third molars will be evaluated for gingival inﬂammation using a modiﬁcation of the Loe and Silness , 1963 GI. The GI uses the following scores: 0 = normal gingiva; 1 = mild inﬂammation; 2 = moderate inﬂammation; and 3 = severe inﬂammation. Gingival index will be evaluated at four sites per tooth
Periodontal parameters- Change in Plaque Index | • At baseline (before 20 weeks gestation) • 8 weeks after completion of periodontal therapy • Within 1-2 days of delivery
  Plaque index (PI). Prebrushing plaque scores for the buccal surface of each tooth will be assigned using a zero to three scale (Silness and Loe, 1964 ) PI, with ''0''indicating an absence of plaque on the clinical crown and a ''3'' indicating the presence of soft deposits covering more than two-thirds of the crown.
  Plaque index will be evaluated at four sites per tooth
Periodontal parameters-Change in Bleeding on probing | • At baseline (before 20 weeks gestation) • 8 weeks after completion of periodontal therapy • Within 1-2 days of delivery
  Bleeding on probing will be evaluated at six sites per tooth
Periodontal parameters- Change in Probing depth (PD) | • At baseline (before 20 weeks gestation) • 8 weeks after completion of periodontal therapy • Within 1-2 days of delivery
  A manual periodontal probe UNC-15, Hu-Friedy, Chicago, IL ,will be used to record on all teeth present in the mouth. Probing depth will be calculated from gingival margin to base of pocket.
  Probing depth will be evaluated at six sites per tooth
Periodontal parameters- Change in Clinical attachment level (CAL) | • At baseline (before 20 weeks gestation) • 8 weeks after completion of periodontal therapy • Within 1-2 days of delivery
  A manual periodontal probe UNC-15, Hu-Friedy, Chicago, IL ,will be used to record on all teeth present in the mouth. CAL will be calculated using the clinically detectable cemento-enamel junction (CEJ) as reference and it will be measured from CEJ to base of pocket.
  Clinical attachment level will be evaluated at six sites per tooth

SECONDARY OUTCOMES:
Serum bio markers -Change in Interleukin-6(IL-6) | • At baseline (before 20 weeks gestation) • 8 weeks after completion of periodontal therapy • Within 1-2 days of delivery
  A 5-ml sample of peripheral venous blood will be collected by vein puncture. The blood samples will be centrifuged at 3000 g for 5 min and the serum will be separated. The serum samples will be frozen in plastic vials at -20ºC until further analyzing. Commercially available ELISA assays will be used to measure concentrations of IL-6 in blood samples, according to the manufacturer's recommendations.
Serum bio markers -Change in Prostaglandin-E2 ( PG-E2) | • At baseline (before 20 weeks gestation) • 8 weeks after completion of periodontal therapy • Within 1-2 days of delivery
  A 5-ml sample of peripheral venous blood will be collected by vein puncture. The blood samples will be centrifuged at 3000 g for 5 min and the serum will be separated. The serum samples will be frozen in plastic vials at -20ºC until further analyzing. Commercially available ELISA assays will be used to measure concentrations of PGE2 in blood samples, according to the manufacturer's recommendations.
Pregnancy Outcomes -Preterm birth neonate | • Within 1-2 days of delivery
  Preterm birth < 37 weeks neonate taken from patients record
Pregnancy Outcomes -Low birth weight neonate | • Within 1-2 days of delivery
  Low birth weight < 2500 gms neonate as taken from patients record

CONTACTS AND LOCATIONS:
Overall Officials: Hezekiah Mosadomi, DMD, Study Chair — Riyadh Colleges of Dentistry and Pharmacy
Locations (1):
- Riyadh Colleges of Dentistry and Pharmacy, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Al-Nozha M, Al-Khadra A, Arafah MR, Al-Maatouq MA, Khalil MZ, Khan NB, Al-Mazrou YY, Al-Marzouki K, Al-Harthi SS, Abdullah M, Al-Shahid MS, Al-Mobeireek A, Nouh MS. Metabolic syndrome in Saudi Arabia. Saudi Med J. 2005 Dec;26(12):1918-25. PMID 16380773
- [Background] Al Qahtani NA, Joseph B, Deepthi A, Vijayakumari BK. Prevalence of chronic periodontitis and its risk determinants among female patients in the Aseer Region of KSA. J Taibah Univ Med Sci. 2017 Mar 3;12(3):241-248. doi: 10.1016/j.jtumed.2016.11.012. eCollection 2017 Jun. PMID 31435246
- [Background] Al-Qurashi FO, Yousef AA, Awary BH. Epidemiological aspects of prematurity in the Eastern region of Saudi Arabia. Saudi Med J. 2016 Apr;37(4):414-9. doi: 10.15537/smj.2016.4.14309. PMID 27052284
- [Background] Athyros VG, Ganotakis ES, Elisaf M, Mikhailidis DP. The prevalence of the metabolic syndrome using the National Cholesterol Educational Program and International Diabetes Federation definitions. Curr Med Res Opin. 2005 Aug;21(8):1157-9. doi: 10.1185/030079905x53333. PMID 16083523
- [Background] Benguigui C, Bongard V, Ruidavets JB, Chamontin B, Sixou M, Ferrieres J, Amar J. Metabolic syndrome, insulin resistance, and periodontitis: a cross-sectional study in a middle-aged French population. J Clin Periodontol. 2010 Jul;37(7):601-8. doi: 10.1111/j.1600-051X.2010.01571.x. Epub 2010 May 13. PMID 20492076
- [Background] Blencowe H, Cousens S, Oestergaard MZ, Chou D, Moller AB, Narwal R, Adler A, Vera Garcia C, Rohde S, Say L, Lawn JE. National, regional, and worldwide estimates of preterm birth rates in the year 2010 with time trends since 1990 for selected countries: a systematic analysis and implications. Lancet. 2012 Jun 9;379(9832):2162-72. doi: 10.1016/S0140-6736(12)60820-4. PMID 22682464
- [Background] Dos Prazeres Tavares H, Dos Santos DC, Abbade JF, Negrato CA, de Campos PA, Calderon IM, Rudge MV. Prevalence of metabolic syndrome in non-diabetic, pregnant Angolan women according to four diagnostic criteria and its effects on adverse perinatal outcomes. Diabetol Metab Syndr. 2016 Mar 22;8:27. doi: 10.1186/s13098-016-0139-3. eCollection 2016. PMID 27006707
- [Background] Green SB. How Many Subjects Does It Take To Do A Regression Analysis. Multivariate Behav Res. 1991 Jul 1;26(3):499-510. doi: 10.1207/s15327906mbr2603_7. PMID 26776715
- [Background] Ide M, Papapanou PN. Epidemiology of association between maternal periodontal disease and adverse pregnancy outcomes--systematic review. J Clin Periodontol. 2013 Apr;40 Suppl 14:S181-94. doi: 10.1111/jcpe.12063. PMID 23627328
- [Background] Iheozor-Ejiofor Z, Middleton P, Esposito M, Glenny AM. Treating periodontal disease for preventing adverse birth outcomes in pregnant women. Cochrane Database Syst Rev. 2017 Jun 12;6(6):CD005297. doi: 10.1002/14651858.CD005297.pub3. PMID 28605006
- [Background] International Diabetes Federation. Information on the IDF consensus worldwide definition of the metabolic syndrome. http://www.idf.org/webdata/docs/IDF_Meta_def_final.pdf Accessed 2014 Apr 10.
- [Background] Knight ET, Liu J, Seymour GJ, Faggion CM Jr, Cullinan MP. Risk factors that may modify the innate and adaptive immune responses in periodontal diseases. Periodontol 2000. 2016 Jun;71(1):22-51. doi: 10.1111/prd.12110. PMID 27045429
- [Background] Fiorini T, Susin C, da Rocha JM, Weidlich P, Vianna P, Moreira CH, Bogo Chies JA, Rosing CK, Oppermann RV. Effect of nonsurgical periodontal therapy on serum and gingival crevicular fluid cytokine levels during pregnancy and postpartum. J Periodontal Res. 2013 Feb;48(1):126-33. doi: 10.1111/j.1600-0765.2012.01513.x. Epub 2012 Jul 27. PMID 22835005
- [Background] Grundy SM. Metabolic syndrome pandemic. Arterioscler Thromb Vasc Biol. 2008 Apr;28(4):629-36. doi: 10.1161/ATVBAHA.107.151092. Epub 2008 Jan 3. PMID 18174459
- [Background] LOE H, SILNESS J. PERIODONTAL DISEASE IN PREGNANCY. I. PREVALENCE AND SEVERITY. Acta Odontol Scand. 1963 Dec;21:533-51. doi: 10.3109/00016356309011240. No abstract available. PMID 14121956
- [Background] Offenbacher S, Beck JD, Jared HL, Mauriello SM, Mendoza LC, Couper DJ, Stewart DD, Murtha AP, Cochran DL, Dudley DJ, Reddy MS, Geurs NC, Hauth JC; Maternal Oral Therapy to Reduce Obstetric Risk (MOTOR) Investigators. Effects of periodontal therapy on rate of preterm delivery: a randomized controlled trial. Obstet Gynecol. 2009 Sep;114(3):551-559. doi: 10.1097/AOG.0b013e3181b1341f. PMID 19701034
- [Background] Page RC, Eke PI. Case definitions for use in population-based surveillance of periodontitis. J Periodontol. 2007 Jul;78(7 Suppl):1387-99. doi: 10.1902/jop.2007.060264. PMID 17608611
- [Background] Penova-Veselinovic B, Keelan JA, Wang CA, Newnham JP, Pennell CE. Changes in inflammatory mediators in gingival crevicular fluid following periodontal disease treatment in pregnancy: relationship to adverse pregnancy outcome. J Reprod Immunol. 2015 Nov;112:1-10. doi: 10.1016/j.jri.2015.05.002. Epub 2015 May 27. PMID 26093363
- [Background] Sanz M, D'Aiuto F, Deanfield J, Fernandez-Avilés F. European workshop in periodontal health and cardiovascular disease-scientific evidence on the association between periodontal and cardiovascular diseases: A review of the literature. Eur Heart J Suppl 2010;12 Suppl B:B3-12
- [Background] SILNESS J, LOE H. PERIODONTAL DISEASE IN PREGNANCY. II. CORRELATION BETWEEN ORAL HYGIENE AND PERIODONTAL CONDTION. Acta Odontol Scand. 1964 Feb;22:121-35. doi: 10.3109/00016356408993968. No abstract available. PMID 14158464